CLINICAL TRIAL: NCT03558659
Title: Positional Therapy to Treat Obstructive Sleep Apnea in Stroke Patients: A Randomized Controlled
Brief Title: Positional Therapy to Treat Obstructive Sleep Apnea in Stroke Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment.
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Mark Boulos, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 122-2018
Record Dates: First submitted 2018-05-23; First posted 2018-06-15 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Stroke, Ischemic; Obstructive Sleep Apnea
Keywords: Stroke; Obstructive sleep apnea; Positional therapy
MeSH Terms: conditions — Ischemic Stroke; Sleep Apnea, Obstructive; Stroke

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positional Therapy Belt (Experimental): Use of positional therapy belt (SlumberBUMP) during sleep.
  Interventions: Device: Positional therapy belt
- Standard Care (No Intervention): No positional therapy belt provided for use during sleep.

INTERVENTIONS:
Device: Positional therapy belt — The positional therapy belt produced by SlumberBUMP will be used by stroke patients during sleep, which helps to avoid sleep in the supine position.
  Other Names: SlumberBUMP positional therapy belt
  Arms: Positional Therapy Belt

SUMMARY:
Obstructive sleep apnea (OSA) has been found to be very common in stroke patients. Obstructive sleep apnea has been found to impede stroke rehabilitation and recovery. However, currently, there are few treatment options for OSA in stroke patients. Continuous positive airway pressure (CPAP) is the current therapy commonly used for OSA in the general population, however stroke patients are not highly compliant with this device. Therefore, we have decided to propose a more feasible alternative to treating obstructive sleep apnea through positional therapy. Positional therapy involves using a device to prevent patients from sleeping on their backs, since this position has been found to exacerbate obstructive sleep apnea. Therefore, we hypothesize that stroke patients who use the positional therapy belt will experience improvements in the severity of OSA.

DETAILED DESCRIPTION:
1. BACKGROUND

   Obstructive sleep apnea is very common in stroke patients, with reported prevalence rates between 30% and 70%. Recent studies suggest that it represents both a risk factor and a consequence of stroke and affects stroke recovery, outcome, and recurrence. A case-control study found that stroke patients with OSA had worse neurological status, lower functional independence scores, and a longer period of hospitalization than stroke patients without OSA. Furthermore, leaving OSA untreated after stroke affects rehabilitation efforts and short- and long-term stroke recovery and outcomes. Current literature supports the implementation of treatment protocols for OSA post-stroke in stroke units. This warrants the need to improve treatment of OSA in stroke patients as a means of secondary prevention and improvement of stroke outcomes.

   1.1 Treating OSA in stroke patients

   Continuous positive airway pressure (CPAP) is the current gold standard therapy for OSA in the general population. Early CPAP therapy was found to have a positive effect on long-term survival in ischaemic stroke patients with moderate-severe OSA. However, CPAP is generally poorly tolerated by stroke patients and has a low compliance. Another alternative therapy, nasal expiratory positive airway pressure (EPAP), was also found to be an ineffective alternative to CPAP in acute stroke patients with OSA.

   Since sleeping in the supine position increases the chance of sleep apnea due to the tendency of the tongue to fall back and block the pharyngeal airway, having stroke patients sleep in a lateral position may improve OSA severity. As sleeping in the supine position is very common in acute stroke patients, positional therapy that reduces supine sleep may be beneficial in treating OSA in stroke patients.

   Positional therapy was found to be as effective as CPAP therapy in patients of the general population with positional OSA and in those patients who are intolerant to CPAP therapy. A pilot RCT found that positional therapy reduced the amount of supine positioning by 36% and AHI was reduced by 19.5% in stroke patients.

   Despite the modest improvements observed from position therapy in stroke patients, there is still a need for a vigorous randomized controlled trial to study the effectiveness of positional therapy to reduce the severity of OSA in stroke patients.
2. RATIONALE

   It is of great importance to routinely diagnose and treat OSA after stroke because OSA is highly prevalent and influences rehabilitation and recovery efforts after stroke. Since CPAP, the current gold standard therapy for OSA, is poorly tolerated by stroke patients and is not conveniently accessible in the hospital, positional therapy for OSA may be a feasible alternative. Positional therapy belts have the advantages of being convenient for patients and may also be economically attractive, however they are not routinely used in Ontario hospital or clinics. Therefore, this warrants the investigation of the effectiveness and feasibility of positional therapy in stroke patients.
3. SIGNIFICANCE

   Our project could substantially change the way healthcare is delivered for stroke patients if it finds that treating OSA with positional therapy improves clinical outcomes after stroke. Since CPAP, the current gold-standard for treating OSA, is poorly tolerated in stroke patients, positional therapy has the potential to provide therapy that is convenient and easy to use for stroke patients. Positional therapy devices can also be easily used in patient hospital beds or homes to treat their OSA. This novel approach would have the potential to improve patient outcomes while reducing healthcare spending and could be easily applied to settings outside of Sunnybrook HSC. Although our study will only examine stroke patients, future work could examine the role of positional therapy in other patient populations. Overall, our study will have an important impact on healthcare delivery and optimizing patient outcomes.
4. RESEARCH OBJECTIVES

The primary objective of our randomized controlled trial is to determine whether positional therapy can effectively treat OSA in patients who have sustained a stroke. This will be evaluated by measuring OSA severity, as assessed by the apnea-hypopnea index (AHI) and oxygen desaturation. AHI and oxygen saturation are both measured using the Resmed ApneaLink device.

The secondary objectives include determining the effectiveness of positional therapy in reducing the time spent in the supine position during sleep. This will be measured using a portable body position sensor, available on the Resmed ApneaLink device. We will also assess if positional therapy improves actigraphy-derived measures (e.g. sleep efficiency and wake after sleep onset) by using Phillips Respironics actigraphy. Furthermore, we seek to explore whether positional therapy improves neurological outcomes (National Institutes of Health Stroke Scale, Montreal Cognitive Assessment, Modified Rankin), psychomotor outcomes (psychomotor vigilance test), psychosocial outcomes (depression, quality of life), performance of daily activities, daytime sleepiness, and length of stay in hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Acute ischemic stroke
2. Patient has been treated at Sunnybrook Health Sciences Centre

Exclusion Criteria:

1. Patients who are unable to lie in a supine position (can be due to existing medical conditions)
2. Patients who are using positive airway pressure therapy or supplemental oxygen at the time of the study
3. Patients who are unable to use the portable sleep monitoring device
4. Physical impairment, aphasia, language barrier, facial/bulbar weakness or trauma restricting the ability to use the portable sleep monitor, and absence of caregiver who can provide assistance
5. Women who are pregnant during the study period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
Change in obstructive sleep apnea severity (Apnea-hypopnea index) | Baseline (within 1 week of study enrollment), follow-up 1 (within 2 weeks of baseline), follow-up 2 (within 3-6 months of baseline)
  Apnea-hypopnea index will be measured using the Resmed ApneaLink device
Change in obstructive sleep apnea severity (oxygen desaturation) | Baseline (within 1 week of study enrollment), follow-up 1 (within 2 weeks of baseline), follow-up 2 (within 3-6 months of baseline)
  Oxygen desaturation will be measured using the Resmed ApneaLink device

SECONDARY OUTCOMES:
Change in time spent in the supine position during sleep | Baseline (within 1 week of study enrollment), follow-up 1 (within 2 weeks of baseline), follow-up 2 (within 3-6 months of baseline)
  Proportion of time spent on supine position during sleep will be measured using a portable body position sensor available on the Resmed ApneaLink device
Change in sleep efficiency (actigraphy) | Baseline (within 1 week of study enrollment), follow-up 1 (within 2 weeks of baseline), follow-up 2 (within 3-6 months of baseline)
  Sleep efficiency will be measured using Phillips Respironics actigraphy
Change in neurological outcomes (National Institutes of Health Stroke Scale) | Baseline (within 1 week of study enrollment), follow-up 1 (within 2 weeks of baseline), follow-up 2 (within 3-6 months of baseline)
  National Institutes of Health Stroke Scale will be used to measure impairment caused by a stroke. The score ranges from 0 to 42, with higher scores meaning greater stroke severity.
Hospital length of stay | Within 3-6 months of baseline
  Hospital length of stay (number of days from time of stroke admission to discharge)
Change in reaction time (psychomotor vigilance test) | Baseline (within 1 week of study enrollment), follow-up 1 (within 2 weeks of baseline), follow-up 2 (within 3-6 months of baseline)
  Psychomotor vigilance will be assessed using a reaction-time test
Change in neurological outcomes (Montreal Cognitive Assessment) | Baseline (within 1 week of study enrollment), follow-up 2 (within 3-6 months of baseline)
  Neurological outcomes (Montreal Cognitive Assessment)
Change in psychological outcomes (Centre for Epidemiological Studies Depression Scale) | Baseline (within 1 week of study enrollment), follow-up 2 (within 3-6 months of baseline)
  Centre for Epidemiological Studies Depression Scale quantifies symptoms related to depression. Scores range from 0 to 60, with higher scores indicating greater depressive symptoms.
Change in quality of life (SF-12 quality of life questionnaire) | Baseline (within 1 week of study enrollment), follow-up 2 (within 3-6 months of baseline)
  SF-12 quality of life questionnaire quantifies quality of life. Scores range from 12 to 47, with low scores indicating poorer quality of life.
Change in daytime sleepiness (Epworth sleepiness scale) | Baseline (within 1 week of study enrollment), follow-up 1 (within 2 weeks of baseline), follow-up 2 (within 3-6 months of baseline)
  Epworth sleepiness scale quantifies daytime sleepiness. Scores range from range from 0 to 24, with higher scores indicating higher average sleep propensity in daily life (daytime sleepiness).
Change in neurological outcomes (Modified Rankin scale) | Baseline (within 1 week of study enrollment), follow-up 2 (within 3-6 months of baseline)
  Modified Rankin scale measures the degree of disability or dependence in the daily activities of people who have suffered a stroke. The scale ranges from 0-6, in which 0 indicates no disability or symptoms and 6 indicating death.
Change in performance in activities of daily living (Barthel Index) | Baseline (within 1 week of study enrollment), follow-up 2 (within 3-6 months of baseline)
  Barthel Index quantifies performance in activities of daily living. The scores range from 0 to 20, with lower scores indicating increased disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wheeler NC, Wing JJ, O'Brien LM, Hughes R, Jacobs T, Claflin E, Chervin RD, Brown DL. Expiratory Positive Airway Pressure for Sleep Apnea after Stroke: A Randomized, Crossover Trial. J Clin Sleep Med. 2016 Sep 15;12(9):1233-8. doi: 10.5664/jcsm.6120. PMID 27306393
- [Background] Wallace DM, Ramos AR, Rundek T. Sleep disorders and stroke. Int J Stroke. 2012 Apr;7(3):231-42. doi: 10.1111/j.1747-4949.2011.00760.x. Epub 2012 Feb 15. PMID 22336145
- [Background] Svatikova A, Chervin RD, Wing JJ, Sanchez BN, Migda EM, Brown DL. Positional therapy in ischemic stroke patients with obstructive sleep apnea. Sleep Med. 2011 Mar;12(3):262-6. doi: 10.1016/j.sleep.2010.12.008. PMID 21306949
- [Background] Srijithesh PR, Aghoram R, Goel A, Dhanya J. Positional therapy for obstructive sleep apnoea. Cochrane Database Syst Rev. 2019 May 1;5(5):CD010990. doi: 10.1002/14651858.CD010990.pub2. PMID 31041813
- [Background] Permut I, Diaz-Abad M, Chatila W, Crocetti J, Gaughan JP, D'Alonzo GE, Krachman SL. Comparison of positional therapy to CPAP in patients with positional obstructive sleep apnea. J Clin Sleep Med. 2010 Jun 15;6(3):238-43. PMID 20572416
- [Background] Parra O, Sanchez-Armengol A, Capote F, Bonnin M, Arboix A, Campos-Rodriguez F, Perez-Ronchel J, Duran-Cantolla J, Martinez-Null C, de la Pena M, Jimenez MC, Masa F, Casadon I, Alonso ML, Macarron JL. Efficacy of continuous positive airway pressure treatment on 5-year survival in patients with ischaemic stroke and obstructive sleep apnea: a randomized controlled trial. J Sleep Res. 2015 Feb;24(1):47-53. doi: 10.1111/jsr.12181. Epub 2014 Jul 21. PMID 25040553
- [Background] Hermann DM, Bassetti CL. Role of sleep-disordered breathing and sleep-wake disturbances for stroke and stroke recovery. Neurology. 2016 Sep 27;87(13):1407-16. doi: 10.1212/WNL.0000000000003037. Epub 2016 Aug 3. PMID 27488603
- [Background] Aaronson JA, van Bennekom CA, Hofman WF, van Bezeij T, van den Aardweg JG, Groet E, Kylstra WA, Schmand B. Obstructive Sleep Apnea is Related to Impaired Cognitive and Functional Status after Stroke. Sleep. 2015 Sep 1;38(9):1431-7. doi: 10.5665/sleep.4984. PMID 25669178